CLINICAL TRIAL: NCT03732404
Title: Effects of Oral Preoperative Carbohydrate on Early Postoperative Outcome After Cesarean Section. A Double-Blind Placebo-controlled Study
Brief Title: Oral Preoperative Carbohydrate on Early Postoperative Outcome After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/197/7/18
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cesarean Section Complications
Keywords: Enhanced recovery after surgery; Preoperative carbohydrate drink; cesarean section

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which was used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative carbohydrate loading (Experimental): Patients in the treatment group will receive a carbohydrate beverage (total carbohydrates equal to 12.6g/100 mL: 2.1 g monosaccharide, 10.0 g maltodextrin; 240 mOsm/L) in a dose of 800 mL. Patients will be free to drink the beverage from the evening before the operation and up to 2 hours before the induction of anesthesia
  Interventions: Drug: preoperative carbohydrate loading
- Placebo (Placebo Comparator): The control group will receive plain water with the same volume and timing of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: preoperative carbohydrate loading — Patients in the treatment group will receive a carbohydrate beverage (total carbohydrates equal to 12.6g/100 mL: 2.1 g monosaccharide, 10.0 g maltodextrin; 240 mOsm/L) in a dose of 800 mL. Patients will be free to drink the beverage from the evening before the operation and up to 2 hours before the induction of anesthesia
  Other Names: Experimental
  Arms: preoperative carbohydrate loading
Drug: Placebo — The control group will receive plain water with the same volume and timing of treatment.
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
Preoperative carbohydrate treatments have been widely adopted as part of enhanced recovery after surgery (ERAS) or fast-track surgery protocols. Although fast-track surgery protocols have been widely investigated and have been shown to be associated with improved postoperative outcomes, some individual constituents of these protocols, including preoperative carbohydrate treatment, have not been subject to such robust analysis.

DETAILED DESCRIPTION:
Carbohydrate (sugar-containing) nutritional supplements have become a routine part of the package of care for people undergoing planned surgical procedures. the investigator wanted to discover whether carbohydrate supplements are a useful part of care packages used by doctors to improve recovery after planned cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing elective caesarean section
* Term gestational age (37+0 to 41+6 weeks)
* Singleton gestation

Exclusion Criteria:

* Women with gestational diabetes and diabetes mellitus
* Fetal intrauterine growth restriction
* Ante-natally detected congenital anomaly which will require admission to the neonatal nursery
* Women who received steroids within the past 7 days prior to delivery
* Women who did not complete a gestational diabetes screening test

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant female scheduled for elective cesarean section
Enrollment: 200 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 3 weeks
  Number of days in the hospital for each participant between the groups.

SECONDARY OUTCOMES:
number of participants experienced nausea | 24 hours postoperative
  Number of participants experienced nausea
Change in preoperative well-being assessment from baseline to one hour using the 100 millimeter (mm) visual analogue scale | ist 24 hours postoperative
  100 mm visual analogue scales for hunger, thirst, anxiety, fatigue and nausea administered on the morning of surgery prior to morning beverage consumption and 60 minutes after the beverage. All measurements will be assessed using the same scale starting at 0 to 100mm with 0 being the worst and 100 being the best and average being 85.
neonatal blood glucose concentration at four and ten hours of age | 24 hours post operative
  measure neonatal blood glucose level at four and ten hours of age
Neonates with plasma glucose level of less than 45 mg/dL between the groups | ist 24 hours postoperative
  First umbilical cord blood sample will be taken for plasma glucose level of less than 45 mg/dL to note hypoglycemia between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided